CLINICAL TRIAL: NCT05845762
Title: Obinutuzumab in the Management of Idiopathic Membranous Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Ying Zhang, Associate chief physician, Qianfoshan Hospital
Other Study IDs: Obinutuzumab-IMN
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — obinutuzumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Response: 1000mg i.v. per day
  Interventions: Drug: Obinutuzumab Injection
- Non-response: 1000mg i.v. per day
  Interventions: Drug: Obinutuzumab Injection

INTERVENTIONS:
Drug: Obinutuzumab Injection — 1000mg intravenous injection
  Other Names: Obinutuzumab

SUMMARY:
To observe the efficacy and safety of obinutuzumab in Chinese population with idiopathic membranous nephropathy and guide clinical management.

DETAILED DESCRIPTION:
Membranous nephropathy (MN) is currently a common histopathological type of adult nephrotic syndrome in China. Its typical feature is the thickening of glomerular basement membrane caused by subepithelial immune complex deposition (mainly IgG and C3). Its prevalence rate in China is increasing year by year, and it has exceeded IgA nephropathy (34.1%) to become the primary glomerular disease with the highest incidence rate. 1. MN can occur at any age and is more common between the ages of 50 and 60. Male to female ratio is 2:1. Primary MN is more common, accounting for about 70%, and secondary MN accounts for about 30%. 40% to 50% of untreated patients with persistent nephrotic syndrome eventually progress to end-stage renal disease (ESRD). The treatment of MN includes symptomatic support therapy without immunosuppressants [controlling blood pressure, lowering urinary protein levels, using angiotensin converting enzyme inhibitors (ACEIs)/angiotensin II receptor blockers (ARBs), etc.] and immunosuppressive therapy. The KDIGO Clinical Practice Guide for Glomerular Diseases in 2021 points out that risk stratification is carried out according to the glomerular filtration rate, serum albumin, urinary protein quantification, anti phospholipase A2 receptor antibody and other indicators of patients, and hormone+cyclophosphamide, hormone+CNIs, or rituximab (CD20 monoclonal antibody) and other treatments are selected according to the degree of risk. In clinical application, alkylating agents have significant toxic side effects, including bone marrow suppression, infection, gonadal suppression, and tumor risk. After 6 to 12 months of treatment with CNIs, 70% to 85% of MN patients can achieve CR or PR. However, the high recurrence rate (40%~50%) is a common problem for patients receiving this regimen, and the risk of chronic nephrotoxicity cannot be underestimated. In recent years, research has found that autoantibodies against the phospholipase A2 receptor (PLA2R) on glomerular podocytes can be detected in most MN patients, while a few patients have antibodies against the platelet reactive protein 7A domain (THSD7A). The possible mechanism is that the antibodies bind to podocyte surface antigens PLA2R or THSD7A, forming immune complexes under glomerular epithelial cells, damaging the glomerular filtration barrier, and subsequently causing proteinuria. These major breakthroughs indicate that primary MN is an autoimmune disease targeting podocytes. The pathogenic role of B cells producing autoantibodies in MN is gradually being recognized, providing strong evidence for the treatment of MN with rituximab (RTX). RTX is a human mouse chimeric monoclonal antibody that specifically targets the surface antigen CD20 of B cells. CD20 is a transmembrane phosphoprotein expressed on the membrane surface of most early and mature B cells. RTX binds to CD20 and consumes CD20+B cells through three ways: antibody dependent cell mediated cytotoxicity, complement dependent cytotoxicity, and direct induction of cell apoptosis. In 2021, the first CD20 monoclonal antibody, rituximab, has been included in the KDIGO guidelines for the clinical treatment of idiopathic membranous nephropathy. However, after seeking medical evidence and clinical work, it has been found that rituximab has a clinical remission rate of 60% in the treatment of idiopathic membranous nephropathy, with about 40% of patients still unresponsive and a high recurrence rate. Researchers are hoping for more treatment options.

Obinutuzumab is a new generation of humanized CD20 monoclonal antibody, which has been confirmed to be stronger than rituximab in vitro B-cell toxicity tests. Otuzumab targets an epitope on CD20 different from that recognized by rituximab, which can cause greater apoptosis of B cells. Modification of the glycan tree structure of the Fc fragment leads to an increase in its affinity for FcgRIII, thus enhancing antibody dependent cytotoxicity through natural killer cell, and enhancing antibody dependent phagocytosis through macrophages. These B cell depletion mechanisms contrast with the main complement dependent cytotoxicity of rituximab. During combined chemotherapy, it has been found that rituximab is more effective in treating certain B-cell malignant tumor patients. Based on these data, altuzumab has become a powerful choice for the new treatment of MN patients. At present, there are only two single center reports abroad with limited data on the experience of treating MN with atozumab, and the results are encouraging. Therefore, the investigators are preparing to conduct a retrospective study on the efficacy of atozumab in the treatment of idiopathic membranous nephropathy at our center, with the aim of providing reference for clinical practice.

3、 Test basis In recent years, the discovery of multiple antibodies has confirmed that idiopathic membranous nephropathy is an autoimmune disease, and the production of autoantibodies by B cells has induced the occurrence of idiopathic membranous nephropathy. The first CD20 monoclonal antibody, rituximab, has been used to treat idiopathic membranous nephropathy and has been included in the 2021 KDOGI guidelines. Otuzumab and rituximab are both CD20, which is different from the human mouse chimerism technique of rituximab. Otuzumab is a fully humanized product, and its mechanism of action is superior to rituximab. Current clinical studies on B lymphocytes have also confirmed the superior therapeutic effect of altuzumab over rituximab, and individual case reports from individual centers have also confirmed the effectiveness of altuzumab in idiopathic membranous nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of nephrotic syndrome.
2. The diagnosis of IMN was confirmed by renal biopsy pathology (light and electron microscopy) or if the serum pla2r antibody was greater than 20 IU / ml.
3. Those who have failed glucocorticoid therapy combined with cyclophosphamide or other immunosuppressive agents or rituximab, or have recurrent relapses.
4. Treatment with inotuzumab.

Exclusion Criteria:

1. Patients with positive HBV serologic markers (HBsAg or / and HBeAg), HCV positivity, or abnormal liver function tests (alt, AST, or bilirubin more than 2 times the upper limit of normal and persistently elevated for 2 weeks).
2. Patients with congenital or acquired immunodeficiency, or combined infections such as active tuberculosis, active CMV, etc. Patients with CO morbid severe infections requiring intravenous antibiotics.
3. Patients with other serious physical or psychological diseases.
4. Patients with congenital heart disease, arrhythmia, heart failure and other severe cardiovascular disease, tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic membranous nephropathy patients receiving obinutuzumab treatment
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Remission | 6 months
  Urine protein quantification was less than 0.3g/24h, renal function was stable and serum albumin was > 35g / L or urinary protein quantification decreased by 50% from baseline and between 0.3-3.5g/24h

IPD SHARING:
Plan to Share IPD: Undecided